CLINICAL TRIAL: NCT04107441
Title: A Phase 1 Ascending Dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Twice Daily Administration of AX-8 Tablets in Healthy Volunteers in a Single-Centre
Brief Title: AX-8 Drug Safety, Tolerability and Plasma Levels in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axalbion SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AX8-002; 2019-002294-57 (EudraCT Number)
Record Dates: First submitted 2019-09-19; First posted 2019-09-27 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: open-label; phase 1; safety; tolerability; pharmacokinetics; healthy volunteers; AX-8

STUDY DESIGN:
Intervention Model Description: A first group of 10 participants will be enrolled in the Part 1 of the study (arm 1).
  Based on the results of Part 1, a second group of 10 participants will be enrolled in Part 2 of the study (arm 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 arm (Experimental): Ten healthy participants will receive one orally disintegrating tablet (ODT) with 5 mg, 10 mg, 20 mg or 40 mg AX-8 twice daily (8 hours apart, i.e. at 0 hour and +8 hours), during the treatment day (Day 1) of treatment periods 1, 2, 3 or 4, respectively.
  Interventions: Drug: AX-8 Part 1
- Part 2 arm (Experimental): Ten healthy participants will receive one orally disintegrating tablet (ODT) with 5 mg AX-8 and one ODT with 40 mg AX-8 8 hours later (i.e. at 0 hour and +8 hours), during the treatment day (Day 1) of the treatment period.
  Interventions: Drug: AX-8 Part 2

INTERVENTIONS:
Drug: AX-8 Part 1 — 5, 10, 20, and 40 mg AX-8 orally disintegrating tablets (ODTs), up to 80 mg/day split over 2 time points, 8 hours apart (i.e. Dose 1: 0 hour and Dose 2: + 8 hours). AX-8 ODTs will be administered orally and will be dissolved on the back of the tongue while the subject is in a sitting position. The subjects will be instructed not to suck, chew or swallow the tablet, i.e. to allow it to dissolve on the back of the tongue without any further intervention.
  Arms: Part 1 arm
Drug: AX-8 Part 2 — 5 and 40 mg AX-8 orally disintegrating tablets (ODTs), 45 mg/day split over 2 time points, 8 hours apart (i.e. Dose 1: 0 hour and Dose 2: + 8 hours). AX-8 ODTs will be administered orally and will be dissolved in the mouth while the subject is in a sitting position. The subjects will be instructed to actively move the tablet around in their mouth (i.e. active oral manipulation of the tablet) until it is fully dissolved.
  Arms: Part 2 arm

SUMMARY:
The main purpose of the study is to see how safe the study drug AX-8 is and how well it is tolerated when administered at different dose levels in healthy participants.

The study will also investigate pharmacokinetics (PK), i.e how the study drug is taken up, metabolized (broken down) and eliminated.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the safety and tolerability of ascending AX-8 oral doses, i.e. orally disintegrating tablets (ODTs), administrated twice for one day (Day 1) in healthy participants.

The secondary objectives are to investigate the pharmacokinetic (PK) profile and the subjective sensory attributes (e.g. basic tastes, palatability, cooling) of ascending AX-8 oral doses (ODTs), administered twice for one day in healthy participants.

The study consists of two parts.

Part 1

The first part of the study (Part 1) is an ascending dose, open-label, single center study in healthy participants. Part 1 will consist of a Screening Period (Days -28 to -1) to assess eligibility to participate in the study, 4 Treatment Periods (Day 1 to Day 2; one overnight stay for each treatment period) with a minimum washout period of 48 hours between doses (however a longer period will be required for dose escalation / safety review decisions, as required) and a Follow-Up Visit 7 to 14 days post last dose.

During each treatment period, participants will be admitted to the study center on the morning of Day 1 and discharged from the study center on the morning of Day 2 (i.e. after the pre-discharge procedures have been performed). Participants will attend a Follow-Up Visit (or Early Withdrawal Visit as applicable) to complete the study.

The end of the study will be the date of the last study visit for the last participant in the study (LPLV).

It is planned to include 10 eligible participants into Part 1 of the study to receive AX-8 ODTs administered orally which will be dissolved on the tongue (oromucosal route of administration). Participants will receive doses of AX-8 ODTs up to 80 mg/day, administered split over 2 dosing time points (i.e. 0 hour and + 8 hours), as follows:

* Treatment Period 1: 2 x 5 mg tablets, 10 mg total;
* Treatment Period 2: 2 x 10 mg tablets, 20 mg total;
* Treatment Period 3: 2 x 20 mg tablets, 40 mg total;
* Treatment Period 4: 2 x 40 mg tablets, 80 mg total.

Dosing in each sequential treatment period will be staggered; after the first 2 participants (i.e. sentinel group) are dosed there will be at least a 24-hour observation period from the morning dose (0 hour) before the remaining 8 participants are dosed. The remaining participants will be dosed if the sentinel group shows no clinically significant safety or tolerability concerns (including available safety electrocardiograms [ECGs], vital signs measurements, physical examinations and review of any adverse events [AEs]) at the discretion of the PI. Any clinically significant findings from the sentinel group in the opinion of the PI will be discussed with the Sponsor prior to dosing of the remaining 8 participants.

Dose escalation will be based on safety and tolerability data from each treatment period. In addition, available PK data from Treatment Period 1 (5 mg; twice daily) and Treatment Period 2 (10 mg; twice daily) will be used to support dose escalation decisions for Treatment Period 3 (20 mg; twice daily) and Treatment Period 4 (40 mg; twice daily).

Escalation to the next higher dose level (i.e. next sequential treatment period) will not take place until the site's PI and the Sponsor have determined that adequate safety and tolerability data from the previous treatment period has been demonstrated to permit proceeding to the next sequential treatment period (i.e. higher dose level). The minimum data package required for dose escalation decisions will include safety and tolerability data through Day 2 in a minimum of 6 participants (including available safety ECGs, vital signs measurements, physical examinations, clinical laboratory tests and review of any adverse events). Safety reports will be produced summarizing the safety data of the participants. The justification for selection of the dose will be prepared by the investigator for the proposed dose escalation and documented in the dose escalation meeting minutes.

Additional participants may be enrolled if it is deemed appropriate by the site's PI and the Sponsor to repeat a dose level or to study an intermediate dose level (lower than those planned). Repetition of a dose level will not be permitted for dose levels that met any of the stopping rules.

Part 2

The first part of the study (Part 1) has been completed, i.e. 10 participants were recruited and received AX-8 (10 mg to 80 mg/day) over 4 treatment periods (in a dose escalation regimen) and have attended their follow-up visits. The interim analysis of the study data from Part 1 has concluded that tablet dissolution time was too long, affecting systemic exposure to AX-8, probably due to the instructions for administration. Consequently, it was decided to re-evaluate the 5 mg and 40 mg AX-8 tablets with other administration instructions.

It is planned that 10 participants will be enrolled into Part 2 of the study to receive a total dose of 45 mg split into two doses on Day 1 (Dose 1 (5 mg): +0 h, Dose 2 (40 mg): + 8 h).

Part 2 will consist of a Screening Period (Days -28 to -1) to assess eligibility to participate in the study, 1 Treatment Period (Day 1 to Day 2; one overnight stay) and a Follow-Up Visit 7 to 14 days post last dose. There will be no dose escalation decisions nor dose staggering of participants as the doses to be administered in Part 2 are lower than the highest dose level administered in Part 1.

For Part 1 and Part 2; blood samples will be taken pre and post each dose to measure plasma concentrations of AX-8, despropyl AX-8 (metabolite C, MetC) and potentially other AX-8 metabolites and compounds. Subjective assessments to characterise the sensory attributes of the AX-8 ODTs (e.g. feeling factors and taste) will be performed pre and post each dose. Safety assessments will be performed throughout the study and will include monitoring adverse events (AEs), physical examinations, vital signs, 12-lead ECGs, and clinical laboratory tests.

The duration of the study will be approximately 65 days for subjects enrolled in Part 1 and approximately 44 days for subjects enrolled in Part 2; however, the actual duration will depend on the length of the screening period and the washout periods (as appropriate).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged ≥ 18 and ≤ 55 years at the time of informed consent
* Female subjects must be either of non-childbearing potential or if of childbearing potential use a highly effective birth control method
* Female subjects (regardless of childbearing potential) must agree not to donate ova/oocytes during the study from the first dosing day and until 30 days after the last dose
* Male subjects with female partners of childbearing potential must be vasectomised with documented medical assessment of the surgical success, or use highly effective contraception together with their female partner(s)
* Male subjects must agree not to donate sperm during the study from the first dosing day and until 90 days after last dose
* Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at Screening
* Have provided written informed consent
* Are willing and able to comply with all aspects of the protocol
* Normal electrocardiogram (ECG) and vital signs (or abnormalities which the clinical Investigator considers the deviation to be irrelevant for the purpose of the study) during screening and prior to first dose
* Laboratory values within the normal range (or the clinical Investigator considers the deviation to be irrelevant for the purpose of the study) during screening
* Findings within the range of clinical acceptability in medical history and physical examination (or the clinical Investigator considers the deviation to be irrelevant for the purpose of the study)

Exclusion Criteria:

* Prior treatment with AX-8
* Hypersensitivity or intolerance to transient receptor potential melastatin subfamily, member 8 (TRPM8) agonists (e.g. menthol, menthol-derivatives, eucalyptol) or any of the excipients of the AX-8 tablets
* Current smoker or individuals who have given up smoking for less than 12 months or ex smoker with > 10 pack-years
* History of upper or lower respiratory tract infection within 4 weeks prior to screening or prior to first dose.
* Requiring concomitant therapy with prohibited medications
* Treatment with biologic therapies within 8 weeks or 5 half-lives, whichever is longer, prior to screening
* Treatment with any investigational therapy within 4 weeks prior to screening
* Serum creatinine, total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > the upper limit of normal (ULN) during screening
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or antibodies against human immunodeficiency virus 1 or 2 (HIV-1 and HIV-2 Abs) during screening
* Positive tests for drugs of abuse or alcohol breath test at screening or prior to first dose
* History of malignancy, with the exception of completely treated and non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin, within 5 years prior to screening
* History of a major psychiatric condition (including major depressive disorder, bipolar disorder, or schizophrenia), suicidal ideation, or suicide attempt
* Presence of any medical condition or disability that, in the Investigator's opinion, could interfere with the assessment of safety or efficacy in this study or compromise the safety of the subject
* History or presence of alcoholism or drug abuse within the past 2 years prior to screening
* Females who are currently pregnant, breastfeeding or lactating, or who have a positive pregnancy test at screening or prior to first dose
* Male subjects with a pregnant, breastfeeding or lactating partner or a partner who is planning to become pregnant during the study or within 90 days after the last dose
* Donation of blood (≥ 400 mL) or plasma, or significant blood loss within 56 days prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Monitoring and recording of AEs will be performed throughout the study.
Changes in biochemistry parameters - Total protein (g/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Albumin (g/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Total bilirubin (μmol/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Alanine transaminase (ALT, IU/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Aspartate transaminase (AST, IU/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Alkaline phosphatase (IU/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Gamma glutamyl transferase (GGT, IU/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Glucose (mmol/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days
  Quantified in participants' plasma.
Changes in biochemistry parameters - Sodium (mmol/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Potassium (mmol/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in biochemistry parameters - Creatinine (μmol/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days
  Quantified in participants' plasma.
Changes in biochemistry parameters - Urea (mmol/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participants' plasma.
Changes in hematology parameters - Hemoglobin (g/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Hematocrit (HTC, %) | From screening visit to follow-up/early withdrawal visit, approximately 65 days
  Quantified in participant's whole blood.
Changes in hematology parameters - Mean cell volume (MCV, fL) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Mean cell hemoglobin (pg) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Mean cell hemoglobin concentration (g/dL) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Platelets (10^9/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Red blood cell count (10^12/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - White blood cell count (10^9/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Absolute neutrophils (10^9/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Absolute lymphocytes (10^9/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Absolute monocytes (10^9/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Absolute eosinophils (10^9/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Absolute basophils (10^9/L) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Percentage neutrophils (%) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Percentage lymphocytes (%) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Percentage monocytes (%) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Percentage eosinophils (%) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in hematology parameters - Percentage basophils (%) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in coagulation parameters - Prothrombin time (PTT, sec) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in coagulation parameters - International normalized ratio (INR) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in coagulation parameters - Activated partial thromboplastin time (aPTT, sec) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Quantified in participant's whole blood.
Changes in urinalysis parameters - Protein (positive or negative) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Glucose (positive or negative) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Specific gravity | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Ketones (positive or negative) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Urobilinogen (normal or abnormal) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Bilirubin (positive or negative) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - pH | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Nitrite (positive or negative) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Leukocytes (positive or negative) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Blood (positive or negative) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - White blood cells (per high power field, HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Red blood cells (HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Bacteria (organisms, HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Hyaline casts (HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Granular casts (HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Cellular casts (HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Epithelial cells (HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in urinalysis parameters - Crystals (HPF) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in vital sign parameters - Body mass index (BMI, kg/m^2) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
  Weight (kg) and height (m) will be combined to report BMI in kg/m^2.
Changes in vital sign parameters - Pulse rate (beats/min) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in vital sign parameters - Systolic blood pressure (mmHg) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in vital sign parameters - Diastolic blood pressure (mmHg) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in vital sign parameters - Tympanic temperature (°C) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in 12-lead electrocardiogram (ECG) parameters - Heart rate (beats/min) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in 12-lead electrocardiogram (ECG) parameters - RR interval (msec) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in 12-lead electrocardiogram (ECG) parameters - PR interval (msec) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in 12-lead electrocardiogram (ECG) parameters - QRS interval (msec) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in 12-lead electrocardiogram (ECG) parameters - QT interval (msec) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.
Changes in 12-lead electrocardiogram (ECG) parameters - QTcF interval (msec) | From screening visit to follow-up/early withdrawal visit, approximately 65 days for Part 1 and 44 days for Part 2.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from the first time point [t=0] to the time point of the last measured concentration [tlast] (AUC0-tlast) of AX-8 and its metabolite (ng.h/mL) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Maximum plasma concentration (Cmax) of AX-8 and its metabolite (ng/mL) for Dose 1 (Cmax1) and Dose 2 (Cmax2) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Percentage area extrapolated to infinity (%AUCx) of AX-8 and its metabolite (ng.h/mL) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Residual area, extrapolated area expressed as fraction of AUC(0-∞) (AUC(t-∞)) of AX-8 and its metabolite (ng.h/mL) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Time of maximum plasma concentration (tmax) of AX-8 and its metabolite for Dose 1 (tmax1) and Dose 2 (tmax2) (h) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Elimination half-life (t½) of AX-8 and its metabolite for Dose 2 only (h) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Elimination rate constant (λz) of AX-8 and its metabolite for Dose 2 only (1/h) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Dose normalized AUC0-tlast: AUC0-tlast / (Dose 1 + Dose 2) of AX-8 and its metabolite (ng.h/mL/mg) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Area under the plasma concentration-time curve from the first time point to the 6th hour (AUC0-6) of AX-8 and its metabolite (ng.h/mL) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Area under the plasma concentration-time curve from the 8th to 14th hour (AUC8-14) of AX-8 and its metabolite (ng.h/mL) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Area under the plasma concentration-time curve from the first time point to the 24th hour (AUC0-24) of AX-8 and its metabolite (ng.h/mL) | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Accumulation based on AUC (RAUC): AUC0-6 / AUC8-14 of AX-8 and its metabolite | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Accumulation based on Cmax (RCmax): Cmax2 / Cmax1 of AX-8 and its metabolite | Part 1 and Part 2: Treatment periods (Days 1 and 2).
Dose normalized Cmax: Cmax1 / Dose 1 of AX-8 and its metabolite | Part 1 and Part 2: Treatment periods (Days 1 and 2).
AX-8 ODT cooling VAS (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Intensity of cooling scored with a 100-mm visual analog scale (VAS) as part of a cooling questionnaire.
AX8-ODT taste and palatability VAS - Sweet taste (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Intensity of sweet taste of the AX-8 ODTs scored with 100-mm visual analog scales (VAS) as part of a taste and palatability questionnaire.
AX8-ODT taste and palatability VAS - Sour taste (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Intensity of sour taste of the AX-8 ODTs scored with 100-mm visual analog scales (VAS) as part of a taste and palatability questionnaire.
AX8-ODT taste and palatability VAS - Salty taste (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Intensity of salty taste of the AX-8 ODTs scored with 100-mm visual analog scales (VAS) as part of a taste and palatability questionnaire.
AX8-ODT taste and palatability VAS - Bitter taste (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Intensity of bitter taste of the AX-8 ODTs scored with 100-mm visual analog scales (VAS) as part of a taste and palatability questionnaire.
AX8-ODT taste and palatability VAS - Umami taste (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Intensity of umami taste of the AX-8 ODTs scored with 100-mm visual analog scales (VAS) as part of a taste and palatability questionnaire.
AX8-ODT taste and palatability VAS - Other taste (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Intensity and nature of other taste of the AX-8 ODTs scored with 100-mm visual analog scales (VAS) as part of a taste and palatability questionnaire.
AX8-ODT taste and palatability VAS - Palatability (mm) | Part 1 and Part 2: Treatment periods (Day 1, i.e. treatment day).
  Palatability of the AX-8 ODTs scored with 100-mm visual analog scales (VAS) as part of a taste and palatability questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit (MEU) Ltd
Locations (1):
- Medicines Evaluation Unit (MEU) Ltd, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No